CLINICAL TRIAL: NCT07220837
Title: Randomized Control Trial (RCT) of Online Learning Module to Advance Research Related to People With Disabilities (D2/R3)
Brief Title: Online Learning Module to Advance Research Related to People With Disabilities
Acronym: D2/R3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-17152; 1UM1TR004400 (NIH)
Record Dates: First submitted 2025-09-18; First posted 2025-10-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Developmental Disability; Intellectual Disability; Disability
Keywords: Bias; Attitudes; Perceptions; Inclusion; Translational Science; Representation
MeSH Terms: conditions — Developmental Disabilities; Intellectual Disability; Behavior

STUDY DESIGN:
Intervention Model Description: Parallel Assignment RCT with block randomization by research team role within each arm:
  * n=65 Principal or Co-investigators
  * n=35 other study personnel (i.e. coordinator, interventionist, etc.) Participating researchers (n=200) will be randomly assigned to either of 2 arms (i.e. Experimental- eLearning module or Control- module on disability data sources). Participants will begin their respective intervention modules after completing the baseline KAP survey.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eLearning module (Experimental): Participants (n=100) will view one interactive 30-minute module aimed at increasing KAP of including PWDs in research.
  Interventions: Other: eLearning module
- Control (Other): Participants (n=100) will view two 15-min modules (total~30 mins) one focusing on disability data sources and the other on the medical/social model of disability. Participants will retake the KAP survey again immediately after completing the 2 modules.
  Interventions: Other: Control

INTERVENTIONS:
Other: eLearning module — * Baseline pre-survey (15 minutes)
  * Baseline learning module (30 minutes)
  * Baseline post-survey (10 minutes)
  * Follow-up survey (3-4 weeks later)
  Components of KAP survey:
  Demographics-research experience/role, disability status, exposure to PWDs, etc. (baseline pre-survey only; e.g. not asked at post follow-up survey) Knowledge-short-answer, clinical scenarios, items focused on historical/legislative context, etc.
  Attitudes-validated "Attitudes to Disability Scale" (ADS) developed by a World Health Organization (WHO) working group Perceptions-questions developed by Prosci's Awareness, Desire, Knowledge, Ability, Reinforcement (ADKAR) framework.
  Arms: eLearning module
Other: Control — Disability Statistics Training (University of New Hampshire Link). Modules identify disability data sources via US surveys and measurement hurdles in disability research:
  A) Module 2/Topic 1 (13m:44s):
  Operationalization of Disability in Surveys- covers the two common operationalization methods, the 6 Question Sequence (6QS) and the Washington Group Short Set (WGSS), and the challenges of collecting disability data
  B) Module 3/Topic 1 (13m:48s):
  Disablement Models- conceptually defines models, such as Nagi's Disablement Model, Work Disability, Verbrugge and Jette, and WHO's Definition.
  Other Names: Disability Statistics Training
  Arms: Control

SUMMARY:
This study will measure the effects of a brief one-time eLearning intervention on researcher Knowledge, Attitudes, and Perceptions (KAP) of including people with disabilities (PWDs) in biomedical & behavioral research. Researchers will be recruited from across the Einstein/Montefiore network, and other medical centers with a focus on CTSAs.

DETAILED DESCRIPTION:
According to the Centers for Disease Control and Prevention (CDC), 1 in 4 adults in the U.S. has a disability, approximately 29% of the overall population. Adults with (vs. without) disabilities have higher rates of obesity (41.6% v. 29.6%), smoking (21.9% v. 10.9%), heart disease (9.6% v. 3.4%), and diabetes (15.9% v. 7.6%), and lower rates of preventive care (e.g., mammograms, cervical cancer screening).

Disability may present as salient to others or be non-visible (e.g., autism, Long COVID). Non-visible disabilities comprise 70-80% of all disabilities; robust data finds stronger negative attitudes towards non-visible (vs. visible) disabilities.

People with Disabilities (PWDs) are under-represented in health research. Reasons include: a) structural elements of research: poorly justified exclusion criteria, PWDs not designated as a vulnerable group, b) access barriers: physical, sensory, literacy; and c) PWDs skepticism due to researcher bias, lack of perceived benefit, focus on cure vs. quality of life. Data on provider attitudes towards people with disabilities (PWDs) is scant.

KAP of barriers and benefits are modifiable roadblocks to including PWDs in research. The research team will develop and test tools to increase researcher motivation and capacity to mitigate perceived barriers. For Aims 1 and 2 of D2/R3, the research team engaged the 10 US sites (Einstein is one) that are Clinical and Translational Science Awards (CTSAs) and Intellectual and Developmental Disabilities Research Centers (IDDRCs) for basic/clinical research and University Centers of Excellence in Developmental Disabilities (UCEDDs).

Timeliness - This study is timely and novel as the perception of disability in research settings has shifted in recent years. Made apparent by the NIHs designation of PWDs as a health disparities population and changes to the Research, Condition, and Disease Categories (RCDCs) (i.e., disability research is now included on the list).

This registration is exclusive to Aim 3 of the D2/R3 study.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=18
* Conducts non-disability focused research (in the past 3 years)
* Conducts (primarily) research with/on adults
* Agree to complete the 1-hour baseline session in one sitting

Exclusion Criteria:

* Participant in Aim1/Aim2 of D2/R3 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Attitudes Towards Disability Scale | Pre-intervention at baseline and 3-4 weeks post intervention
  16 item scale - Attitudes to disability scale (ADS). Scoring range on a 5-point Likert scale ranging from 1-5, yielding an overall possible scoring range of 16-80. Participants for whom a single item is inapplicable (i.e., N/A) will have data removed for that item. Lower scores indicate less favorable attitudes towards people with disabilities, while higher scores indicate more favorable attitudes.
  *Note: Questions 1-6 & 11-16 are reverse coded.

SECONDARY OUTCOMES:
Change in Knowledge Scores | Pre-intervention at baseline and 3-4 weeks post intervention
  10 item scale - Changes in Knowledge scores from baseline. Scoring range: 0%-100%, whereby the percentage correct indicates comprehension towards factual items and best practices for engaging people with disabilities. Questions 4, 8, and 10 can be scored for partial credit. Percentage correct scores will be summarized by study arm.
Change in Perception Scores | Pre-intervention at baseline, and 3-4 weeks post intervention
  18 item scale - Change in Perception scores from baseline. Scores are based on 5 domains (i.e. Awareness, Desire, Knowledge, Ability, Reinforcement). Scoring range for each domain includes: Awareness (1-5), Desire (2-10), Knowledge (2-20), Ability (2-20), Reinforcement (6-30). An overall composite score of 13-85 for all 5 of these domains. Participants for whom a single item is inapplicable (i.e., N/A) will have data removed for that item. Higher scores indicate greater Awareness of, desire to, Knowledge about, Ability to, and Reinforcements regarding inclusion of people with disabilities in research.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Bonuck, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
After results are reported in a peer-reviewed manuscript on the trial outcomes all data (i.e. metadata, documentation, protocols, measures) will be shared and associated with the datasets.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: De-identified survey data will be exported from Einstein-Montefiore's REDCap database into a common and open format (e.g., .CSV with variable labels). The survey will have previously been made publicly available in a peer review manuscript including information about our research process, details of the data analysis plan, protocols, etc.
  All dataset(s) that can be shared will be deposited into the Harvard Dataverse Repository (HDR).
Access Criteria: Prior to sharing we will remove all personal identifiers. Survey data will be made available in csv. and will not require specialized tools to gain access or be manipulated (i.e. no restrictions).
  Resources (e.g. code) will be made publicly available through the HDR.
URL: https://support.dataverse.harvard.edu/

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Disability and Health Data System (DHDS). In:2023.
- [Background] Granjon M, Pillaud N, Popa-Roch M, Aubé B, Rohmer O. Attitudes towards invisible disabilities: Evidence from behavioral tendencies. Current Research in Behavioral Sciences. 2025;8:100164.
- [Background] Bonuck K, Fishman A. Reducing translational science roadblocks to disability research. J Clin Transl Sci. 2025 Jun 9;9(1):e174. doi: 10.1017/cts.2025.10073. eCollection 2025. PMID 40979104
- [Background] Havercamp SM, Krahn GL, Larson SA, Fujiura G, Goode TD, Kornblau BL; National Health Surveillance for IDD Workgroup. Identifying People With Intellectual and Developmental Disabilities in National Population Surveys. Intellect Dev Disabil. 2019 Oct;57(5):376-389. doi: 10.1352/1934-9556-57.5.376. PMID 31568737
- [Background] Schieve LA, Gonzalez V, Boulet SL, Visser SN, Rice CE, Van Naarden Braun K, Boyle CA. Concurrent medical conditions and health care use and needs among children with learning and behavioral developmental disabilities, National Health Interview Survey, 2006-2010. Res Dev Disabil. 2012 Mar-Apr;33(2):467-76. doi: 10.1016/j.ridd.2011.10.008. Epub 2011 Nov 24. PMID 22119694
- [Background] Maenner MJ, Shaw KA, Bakian AV, Bilder DA, Durkin MS, Esler A, Furnier SM, Hallas L, Hall-Lande J, Hudson A, Hughes MM, Patrick M, Pierce K, Poynter JN, Salinas A, Shenouda J, Vehorn A, Warren Z, Constantino JN, DiRienzo M, Fitzgerald RT, Grzybowski A, Spivey MH, Pettygrove S, Zahorodny W, Ali A, Andrews JG, Baroud T, Gutierrez J, Hewitt A, Lee LC, Lopez M, Mancilla KC, McArthur D, Schwenk YD, Washington A, Williams S, Cogswell ME. Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2018. MMWR Surveill Summ. 2021 Dec 3;70(11):1-16. doi: 10.15585/mmwr.ss7011a1. PMID 34855725
- [Background] Zablotsky B, Black LI, Maenner MJ, Schieve LA, Danielson ML, Bitsko RH, Blumberg SJ, Kogan MD, Boyle CA. Prevalence and Trends of Developmental Disabilities among Children in the United States: 2009-2017. Pediatrics. 2019 Oct;144(4):e20190811. doi: 10.1542/peds.2019-0811. PMID 31558576
- [Background] Karpur A, Vasudevan V, Shih A, Frazier T. Brief Report: Impact of COVID-19 in Individuals with Autism Spectrum Disorders: Analysis of a National Private Claims Insurance Database. J Autism Dev Disord. 2022 May;52(5):2350-2356. doi: 10.1007/s10803-021-05100-x. Epub 2021 May 26. PMID 34041682
- [Background] McDermott S, Royer J, Cope T, Lindgren S, Momany E, Lee JC, McDuffie MJ, Lauer E, Kurtz S, Armour BS. Using Medicaid Data to Characterize Persons With Intellectual and Developmental Disabilities in Five U.S. States. Am J Intellect Dev Disabil. 2018 Jul;123(4):371-381. doi: 10.1352/1944-7558-123.4.371. PMID 29949427
- [Background] Fujiura GT, Li H, Magana S. Health Services Use and Costs for Americans With Intellectual and Developmental Disabilities: A National Analysis. Intellect Dev Disabil. 2018 Apr;56(2):101-118. doi: 10.1352/1934-9556-56.2.101. PMID 29584559
- [Background] Barth S LS, Simmons T,. Medicaid Services for People with Intellectual or Developmental Disabilities - Evolution of Addressing Service Needs and Preferences 2020.
- [Background] Centers for Disease Control and Prevention, National Center on Birth Defects and Developmental Disabilities, Disability. Disability and Health Data System (DHDS) Data . Centers for Disease Control and Prevention; 2021.
- [Background] Rios D, Magasi S, Novak C, Harniss M. Conducting Accessible Research: Including People With Disabilities in Public Health, Epidemiological, and Outcomes Studies. Am J Public Health. 2016 Dec;106(12):2137-2144. doi: 10.2105/AJPH.2016.303448. Epub 2016 Oct 13. PMID 27736212
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Population Health and Public Health Practice; Committee on Community-Based Solutions to Promote Health Equity in the United States; Baciu A, Negussie Y, Geller A, Weinstein JN, editors. Communities in Action: Pathways to Health Equity. Washington (DC): National Academies Press (US); 2017 Jan 11. Available from http://www.ncbi.nlm.nih.gov/books/NBK425848/ PMID 28418632
- [Background] Swenor B, Deal JA. Disability Inclusion as a Key Component of Research Study Diversity. N Engl J Med. 2022 Jan 20;386(3):205-207. doi: 10.1056/NEJMp2115475. Epub 2022 Jan 15. No abstract available. PMID 35029848
- See also: Eunice Kennedy Shriver National Institute of Child Health and Human Development. A to Z Fact sheets: intellectual and developmental disabilities (IDDs) — https://www.nichd.nih.gov/health/topics/factsheets/idds
- See also: National Institute of Health. (2023, September 26). NIH designates people with disabilities as a population with health disparities. News Releases — https://www.nih.gov/news-events/news-releases/nih-designates-people-disabilities-population-health-disparities
- See also: Centers for Disease Control and Prevention. (2015, April 14). Disability Impacts All of Us Infographic. CDC Disability and Health. — https://www.cdc.gov/disability-and-health/articles-documents/disability-impacts-all-of-us-infographic.html